CLINICAL TRIAL: NCT01034319
Title: Genetic Counseling and Lifestyle Change for Diabetes Prevention
Acronym: GC/LC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Richard W Grant MD MPH, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21DK084527 (NIH); R21DK084527 (NIH)
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Pre-diabetes; Overweight; Metabolic Syndrome
Keywords: type 2 diabetes; genetics; genetic counseling; diabetes prevention
MeSH Terms: conditions — Glucose Intolerance; Overweight; Metabolic Syndrome; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diabetes Genetic Counseling (Experimental): Subjects will have been genotyped and will received genetic counseling based on their results
  Interventions: Behavioral: Diabetes Genetic Counseling
- No Genotyping or Counseling (Placebo Comparator): Patients will not be genotyped and will therefore not receive genetic counseling
  Interventions: Behavioral: No genetic counseling

INTERVENTIONS:
Behavioral: Diabetes Genetic Counseling — Subjects will be genotyped based on a 37-allele aggregate score and counseled regarding the implications of the results prior to enrollment in a 12-week diabetes prevention program
  Arms: Diabetes Genetic Counseling
Behavioral: No genetic counseling — These subjects will not be genotyped or counseled prior to enrollment in a 12-week diabetes prevention program
  Arms: No Genotyping or Counseling

SUMMARY:
This study will examine the impact diabetes genetic counseling on patient motivation and disease prevention behaviors among subjects with pre-diabetes. Intervention subjects will be provided with their individual diabetes genotype risk score derived from aggregating the combined results of 37 diabetes risk-associated genetic loci. Controls will not be tested. All subjects will be enrolled in a 12-week diabetes prevention program.

DETAILED DESCRIPTION:
This study will examine the impact diabetes genetic counseling on patient motivation and disease prevention behaviors among subjects with pre-diabetes. We will randomize subjects with pre-diabetes to genetic testing vs. no genetic testing in order to obtain an unconfounded test of the hypothesis that genetic testing will change patient behavior. Intervention subjects will be provided with their individual diabetes genotype risk score derived from aggregating the combined results of 37 diabetes risk-associated genetic loci. Because patients can receive either "Higher risk" or "Lower risk" genetic test results, we will separately examine the impact of "Higher risk" and "Lower risk" test results compared to untested controls. All subjects will be enrolled in a 12-week diabetes prevention program.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (Body mass index ≥ 29.1 kg/m2 in men, ≥ 27.2 kg/m2 in women) with at least 2 other formal criteria for Metabolic Syndrome (see Table -NCEP ATP-III Criteria)
* Adult (> 21 years of age)
* No diagnosis or treatment for diabetes (Type 1 or Type 2) or cardiovascular disease (e.g. myocardial infraction, coronary bypass surgery, congestive heart failure, peripheral vascular disease)
* Physically able and willing to participate in a 12-week group session curriculum for weight loss and dietary change
* Able to understand and communicate effectively in English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-08 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
stage of change | baseline, after counseling, after completing program (3 months)

SECONDARY OUTCOMES:
program attendance | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Grant, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Practice Based Research Network, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Grant RW, O'Brien KE, Waxler JL, Vassy JL, Delahanty LM, Bissett LG, Green RC, Stember KG, Guiducci C, Park ER, Florez JC, Meigs JB. Personalized genetic risk counseling to motivate diabetes prevention: a randomized trial. Diabetes Care. 2013 Jan;36(1):13-9. doi: 10.2337/dc12-0884. Epub 2012 Aug 28. PMID 22933432
- [Derived] Waxler JL, O'Brien KE, Delahanty LM, Meigs JB, Florez JC, Park ER, Pober BR, Grant RW. Genetic counseling as a tool for type 2 diabetes prevention: a genetic counseling framework for common polygenetic disorders. J Genet Couns. 2012 Oct;21(5):684-91. doi: 10.1007/s10897-012-9486-x. PMID 22302620